CLINICAL TRIAL: NCT05766826
Title: Scaling up Coupons for Safe Water Treatment in Kenya
Brief Title: Coupons for Safe Water Project
Acronym: Coupons
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Abdul Latif Jameel Poverty Action Lab (Other); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DILChlorine Coupons Project
Record Dates: First submitted 2023-02-02; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Death; Death, Infant; Diarrhea; Diarrhea, Infantile; Water-Borne Infectious Disease; Water-Related Diseases
Keywords: Child health; Child mortality; Chlorine; Safe water; Targeting; Coupons; RCT; East Africa; Kenya
MeSH Terms: conditions — Death; Infant Death; Diarrhea; Diarrhea, Infantile; Waterborne Diseases

STUDY DESIGN:
Intervention Model Description: This study will conduct individual randomization, assigning half of the women to receive coupons and the other half to the control group as we enroll.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): After enrollment over a phone call, they receive a SMS text message with an ID number to receive their coupons at the health facility. Those coupons can be used to redeem WaterGuard 150mL dilute chlorine. Participants in this group will receive a packet of coupons that ensure a monthly supply of a150ml bottle of dilute chlorine solution for at least the next 12 months. These coupons are redeemable in health facilities and other sites registered for the study.
  Interventions: Other: Coupons for safe water program: Treatment
- Control Arm (Experimental): After enrollment over a phone call, they will not be contacted.
  Interventions: Other: Coupons for safe water program: Control

INTERVENTIONS:
Other: Coupons for safe water program: Treatment — Randomly selected women in the treatment group will receive coupons for free chlorine solutions to be redeemed at the health facility each month.
  Arms: Treatment Arm
Other: Coupons for safe water program: Control — Randomly selected women in the treatment group will not receive coupons for free chlorine solutions after enrollment.
  Arms: Control Arm

SUMMARY:
Guaranteeing access to safe drinking water is still a challenge in rural households in developing countries, and unsafe water sources are responsible for millions of deaths each year around the world. Coupons for free dilute chlorine solution are a cost-effective and effective way of ameliorating child health and reducing diarrhea incidence. It is still an empirical challenge, however, to see if the positive health effects will be maintained when the program is implemented at scale. In this study, investigators conduct a randomized controlled trial (RCT) at scale to study the impacts of a chlorine coupon program implemented at health clinics on child health, including self-reported diarrhea, fever, and cough incidence in the previous two weeks. Investigators further investigate the pathway of the impact, such as self-reported and objectively measured use of chlorine and frequency of visits to health clinics.

DETAILED DESCRIPTION:
Guaranteeing access to safe drinking water is still a challenge in rural households in developing countries, and unsafe water sources are responsible for millions of deaths each year around the world. Coupons for free dilute chlorine solution are (i) a cost-effective solution to targeting water treatment for households that need it and will use it and (ii) an effective way of ameliorating child health and reducing diarrhea incidence. It is still an empirical challenge, however, to see if the positive health effects will be maintained when the program is implemented at scale. In this study, investigators conduct a randomized controlled trial (RCT) at scale to study the impacts of a chlorine coupon program implemented at health clinics on child health, including self-reported diarrhea, fever, and cough incidence in the previous two weeks. Investigators further study the pathway of the impact, such as self-reported and objectively measured use of chlorine and frequency of visits to health clinics. Investigators monitor the program's impact at Health and Demographic Surveillance Systems (HDSS) sites in collaboration with the Kenya Medical Research Institute (KEMRI). Data collection includes child mortality, as well as verbal autopsies for deceased children. Data on mortality will be useful for future meta-analyses that pool data from multiple studies in order to estimate the mortality impact of free chlorine distribution schemes.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant women
* Women living inside Health and Demographic Surveillance Systems (HDSS) catchment areas.

Exclusion Criteria:

- Women who do not consent.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The recruitment takes place at health facility targeting women visiting health facilities for antenatal care, postnatal care, and other reasons. This study recruits currently pregnant women.
Enrollment: 3468 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Verified chlorine usage - 6 months | The study will measure the presence of free chlorine residual in drinking water 6 months after the program launch.
  Presence of free chlorine residual in the drinking water, as observed through water testing using chlorine test strips. Households with a non-zero concentration of residual chlorine are considered to have treated their water.
Verified chlorine usage - 12 months | The study will measure the presence of free chlorine residual in drinking water 12 months after the program launch.
  Presence of free chlorine residual in the drinking water, as observed through water testing using chlorine test strips. Households with a non-zero concentration of residual chlorine are considered to have treated their water.
Verified chlorine usage - 18 months | The study will measure the presence of free chlorine residual in drinking water 18 months after the program launch.
  Presence of free chlorine residual in the drinking water, as observed through water testing using chlorine test strips. Households with a non-zero concentration of residual chlorine are considered to have treated their water.
Verified chlorine usage - 24 months | The study will measure the presence of free chlorine residual in drinking water 24 months after the program launch.
  Presence of free chlorine residual in the drinking water, as observed through water testing using chlorine test strips. Households with a non-zero concentration of residual chlorine are considered to have treated their water.
Verified chlorine usage - 30 months | The study will measure the presence of free chlorine residual in drinking water 30 months after the program launch.
  Presence of free chlorine residual in the drinking water, as observed through water testing using chlorine test strips. Households with a non-zero concentration of residual chlorine are considered to have treated their water.
Verified chlorine usage - 36 months | The study will measure the presence of free chlorine residual in drinking water 36 months after the program launch.
  Presence of free chlorine residual in the drinking water, as observed through water testing using chlorine test strips. Households with a non-zero concentration of residual chlorine are considered to have treated their water.

SECONDARY OUTCOMES:
Child morbidity - 6 months | The study assesses child morbidity 6 months after the program launch.
  Child morbidity will include caregiver-reported diarrhea, fever, and cough incidents and cost related to sickness in the previous two weeks. This study will be underpowered to detect impacts on mortality, but investigators will collect data on mortality in any case as this study will contribute to a meta-analysis conducted in the future.
Child morbidity - 12 months | The study assesses child morbidity 12 months after the program launch.
  Child morbidity will include caregiver-reported diarrhea, fever, and cough incidents and cost related to sickness in the previous two weeks. This study will be underpowered to detect impacts on mortality, but investigators will collect data on mortality in any case as this study will contribute to a meta-analysis conducted in the future.
Child morbidity - 18 months | The study assesses child morbidity 18 months after the program launch.
  Child morbidity will include caregiver-reported diarrhea, fever, and cough incidents and cost related to sickness in the previous two weeks. This study will be underpowered to detect impacts on mortality, but investigators will collect data on mortality in any case as this study will contribute to a meta-analysis conducted in the future.
Child morbidity - 24 months | The study assesses child morbidity 24 months after the program launch.
  Child morbidity will include caregiver-reported diarrhea, fever, and cough incidents and cost related to sickness in the previous two weeks. This study will be underpowered to detect impacts on mortality, but investigators will collect data on mortality in any case as this study will contribute to a meta-analysis conducted in the future.
Child morbidity - 30 months | The study assesses child morbidity 30 months after the program launch.
  Child morbidity will include caregiver-reported diarrhea, fever, and cough incidents and cost related to sickness in the previous two weeks. This study will be underpowered to detect impacts on mortality, but investigators will collect data on mortality in any case as this study will contribute to a meta-analysis conducted in the future.
Child morbidity - 36 months | The study assesses child morbidity 36 months after the program launch.
  Child morbidity will include caregiver-reported diarrhea, fever, and cough incidents and cost related to sickness in the previous two weeks. This study will be underpowered to detect impacts on mortality, but investigators will collect data on mortality in any case as this study will contribute to a meta-analysis conducted in the future.
Self-reported health facility attendance - 6 months | The study assesses the self-reported health facility attendance 6 months after the program launch.
  Participants will be surveyed about recent visits to health facilities. For women who are currently pregnant or delivered a baby in the last 12 months, the study asks the number of antenatal care visits. For women who have children under age 5, we collect data on the number of postnatal care.
Self-reported health facility attendance - 12 months | The study assesses the self-reported health facility attendance 12 months after the program launch.
  Participants will be surveyed about recent visits to health facilities. For women who are currently pregnant or delivered a baby in the last 12 months, the study asks the number of antenatal care visits. For women who have children under age 5, we collect data on the number of postnatal care.
Self-reported health facility attendance - 18 months | The study assesses the self-reported health facility attendance 18 months after the program launch.
  Participants will be surveyed about recent visits to health facilities. For women who are currently pregnant or delivered a baby in the last 12 months, the study asks the number of antenatal care visits. For women who have children under age 5, we collect data on the number of postnatal care.
Self-reported health facility attendance - 24 months | The study assesses the self-reported health facility attendance 24 months after the program launch.
  Participants will be surveyed about recent visits to health facilities. For women who are currently pregnant or delivered a baby in the last 12 months, the study asks the number of antenatal care visits. For women who have children under age 5, we collect data on the number of postnatal care.
Self-reported health facility attendance - 30 months | The study assesses the self-reported health facility attendance 30 months after the program launch.
  Participants will be surveyed about recent visits to health facilities. For women who are currently pregnant or delivered a baby in the last 12 months, the study asks the number of antenatal care visits. For women who have children under age 5, we collect data on the number of postnatal care.
Self-reported health facility attendance - 36 months | The study assesses the self-reported health facility attendance 36 months after the program launch.
  Participants will be surveyed about recent visits to health facilities. For women who are currently pregnant or delivered a baby in the last 12 months, the study asks the number of antenatal care visits. For women who have children under age 5, we collect data on the number of postnatal care.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kremer, PhD, Principal Investigator — University of Chicago; Pascaline Dupas, PhD, Principal Investigator — Stanford University; Elisa M Maffioli, PhD, Principal Investigator — University of Michigan; Akito Kamei, PhD, Principal Investigator — University of Chicago; Sammy Khagayi, PhD, Principal Investigator — Kenya Medical Research Institute
Locations (2):
- Kenya (2):
  - Health and Demographic Surveillance System (HDSS sites), Kisumu
  - Health and Demographic Surveillance System (HDSS) sites, Siaya

IPD SHARING:
Plan to Share IPD: Yes
Once the analysis is complete, the de-identified data will be deposited in the public server for replicability of the research analysis.
Time Frame: After the completion of the whole study
Access Criteria: The de-identified data will be deposited in the public server